CLINICAL TRIAL: NCT06429839
Title: Nimotuzumab Concurrent With Chemoradiotherapy for Elderly or Malnourished Patients With Unresectable Esophageal Squamous Cell Carcinoma: A Phase II Study
Brief Title: Nimotuzumab Concurrent With Chemoradiotherapy for Esophageal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4571
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer; Nimotuzumab; Chemoradiotherapy; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nimotuzumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab concurrent with chemordiotherapy followed by surgery (Experimental)
  Interventions: Combination Product: Nimotuzumab with chemoradiotherapy

INTERVENTIONS:
Combination Product: Nimotuzumab with chemoradiotherapy — Radiotherapy,40-50.4Gy/20-28f. Nimotuzumab 400mg,ivgtt,W2d. Chemotherapy, S-1,40-60mg/m2, on BSA, orally twice daily on radiotherapy days.

SUMMARY:
Elderly or malnourished patients diagnosed with locally advanced esophageal squamous cell carcinoma (ESCC) had poor prognosis. Radiotherpy was an important and effective treatment in treating ESCC. The present study is a one-arm trial that seeks to evaluate the efficacy in patients with unresectable ESCC. The study objectives include R0 resection rate, complete pathological response and treatment toxicity, etc.

Nimotuzumab is a recombinant humanized monoclonal antibody against EGFR. Its efficacy and safety in patients with esophageal cancer have been confirmed by many studies.

The current prospective phase II study aimed to evaluate the efficacy and safety of a combination regimen comprising chemotherapy with nimotuzumab with a dose of 800mg per week and S-1 and concurrent radiotherapy for patients who are elderly or malnourished.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma.
* No previous treatment for the esophageal carcinoma.
* KPS score ≥70.
* NRS-2002 score≥2.
* Main organs and bone marrow function are normal: routine blood tests: hemoglobin (Hb) ≥100g/L ; absolute neutrophil count (NEUT)≥1.5×109/L; platelets (PLT) ≥100×109/L; white blood cell (WBC)≥3.5×109/L,biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×UNL; serum total bilirubin (TBIL) ≤1.5×UNL; serum creatinine ( Cr) 1.0×1.5UNL, and BUN≤1.0×UNL;

Exclusion Criteria:

* Previous treatment of the esophageal cancer with surgery, radiation, or chemotherapy.
* Those combined with other primary malignant tumors other than esophageal cancer (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* At the time of diagnosis, there were distant and hematogenous metastases beyond the supraclavicular lymph node region, including retroperitoneal multiple lymph node metastasis, bone metastasis, brain metastasis, lung metastasis, liver metastasis, malignant pleural effusion and ascites
* There are active infections, such as active tuberculosis and hepatitis
* There are contraindications to targeted therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 4 months after initiation of induction chemoimmunotherapy
  Minimal distance tumor/circumferential resection margin (CRM) > 1 mm.

SECONDARY OUTCOMES:
Pathological complete response | 4 months after initiation of induction chemoimmunotherapy
  the complete remission of all viable cancer cells in any of the specimens from surgery, including the primary site and lymph nodes
Event-free survival | 1 month after chemoradiotherapy
  the time from start of chemoradiotherapy to 1 month after chemoradiotherapy
Postoperative complications | 1 month after surgery
Overall survival | 1 year after all treatment
  the time from start of induction chemo(immuno)therapy to all-cause death, or the last day of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China